CLINICAL TRIAL: NCT03137316
Title: Prevalence of Secondary Hyperparathyroidism Among Patients With Diabetic Nephropathy
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Collaborators: New Jeddah Clinic Hospital (Industry)
Responsible Party: Principal Investigator, Mahmoud Hamada imam, Lecturer in Internal Medidicne Department- Faculty of Medicine, Benha University
Other Study IDs: BN-0418
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Secondary Hyperparathyroidism; Diabetic Nephropathies
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: intact parathyroid hormone level — obtain intact parathyroid hormone level from patients records.

SUMMARY:
The aim of this study is to evaluate the prevalence of secondary hyperparathyroidism among patients with diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* [1] Age was above 18 years, [2] Patient had diabetic nephropathy which was diagnosed based on the presence of urinary albumin/creatinine ratio (uACR) ≥ 30 mg/gm ± 24 hours' urinary protein measurement ≥ 300 mg/day

Exclusion Criteria:

* [1] patients were already receiving cinacalcet and/or [2] patients had undergone neck surgery for parathyroidectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 437 diabetic patients were enrolled in this study from 864 diabetic patients who attended diabetes and nephrology outpatient clinics in our tertiary care hospital in Jeddah from Jan 2014 to Feb 2017.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
intact parathyroid level | within 1 hour from attending in the clinic
  intact parathyroid level

IPD SHARING:
Plan to Share IPD: No